CLINICAL TRIAL: NCT04622189
Title: Neuro-rehabilitation of Upper Limb Stroke Patients Through Motor Resonance and Mirror Neurons
Brief Title: Action Observation Training for Upper Limb Rehabilitation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Istituto Italiano di Tecnologia (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, PhD, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brain_AOT_stroke
Record Dates: First submitted 2020-10-29; First posted 2020-11-09 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Stroke Rehabilitation
Keywords: Stroke; Rehabilitation; AOT; kinematic; brain plasticity; mirror neuron system
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Action observation training for the upper limb rehabilitation (Experimental): Neurorehabilitation training for the upper limb using AOT consists of watching videos related to every day actions. The subjects will be asked to reproduce, as accurately as possible, the actions proposed by the system, that will record their execution. In order to keep high motivation and participation in activities, simple games of skill will also be created that will involve the patient on both the motor and cognitive side. The training program includes 250 videos of every day transitive and intransitive actions: 20 consecutive sessions of 1 hour, five times a week over four weeks.
  Interventions: Device: Action observation training

INTERVENTIONS:
Device: Action observation training — Integration of four main tools:
  * PATIENT INTERFACE, which has been implemented to present stimuli with a user friendly interface, with personalized menu and with the possibility to manage the training program; user personal page containing user information and history of activities with daily performance are stored too.
  * MOCAP during action imitation will be recorded using MindMotion infrared camera to capture the trunk movement while an electromagnetic system (Trackstar from NDI) will be used to record fingers fine movements.
  * EEG data will be collected during video observation using an Enobio wireless system integrated with the platform.

SUMMARY:
The purpose of this study is to assess the changes in physiological parameters and clinical scales resulting from treatment with AOT (action observation training) in subjects with subacute stroke. Furthermore, this study assess the perception of applicability and satisfaction degree for this kind of treatments.

DETAILED DESCRIPTION:
After being informed about the study, all patients give written informed consent and will undergo a 1-week screening period to determine eligibility for study entry. Patient who meet the eligibility requirements will be given clinical and instrumental assessments before the start of treatment (T0) after 3 weeks (T1), at the end of the treatment (T2) and after 6 months (T3). A training program of 4 weeks including 250 videos of every day actions has been developed. Videos includes transitive and intransitive actions. Each week has a five day program, each day is divided in three sessions, in each session there are observation and imitation and attentional questions. AOT is always performed in conjunction with the conventional rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Should had experienced first ever ischemic or haemorrhagic stroke
* Fugl-Meyer Assessment < 55
* normal or corrected to normal visual acuity

Exclusion Criteria:

* presence of severe neuropsychological disorders
* medical conditions likely to interfere with the ability to safely complete the study protocol
* pain in the upper limb assessed with the Visual Analogue Scale (VAS)> 7
* intracranial metal implants
* history of seizures or epilepsy
* severe cardiopulmonary, renal, and hepatic diseases
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment Upper Extremity between four time points | Baseline, week 3, week 4, after 6 months
  Scale that assess the sensorimotor impairment in individuals who have had stroke.
Change in Barthel Index between four time points | Baseline, week 3, week 4,after 6 months
  Scale that measures disability or dependence in activities of daily living in stroke patients.
Change in Box and Block Test between four time points | Baseline, week 3, week 4,after 6 months
  To assess unilateral gross manual dexterity
Change in Modified Ashworth Scale between four time points | Baseline, week 3, week 4,after 6 months
  To measure spasticity. It consists of a 5-point nominal scale using subjective clinical assessments of tone ranging from 0 - 'No increases in tone' to 4 - 'Limb rigid in flexion or extension [abduction/adduction]'. An additional grade is added (1+) for the MAS to indicate resistance in the movement.
Change in Visual Analogue Scale between four time points | Baseline , week 3, week 4,after 6 months
  Scale that consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The length of the line is 10-cm. Measurements from the starting point (left end) of the scale to the patients' marks are recorded in centimeters and are interpreted as their pain.
Electroencephalography power in alpha band | Up to 1 month
  EEG data will be recorded to test presence of particular changes in brain activity in during AOT training. In particular plasticity and mu rhythm desynchronization will be investigated.
Motion Capture (MOCAP) recordings | Up to 1 month
  Kinematic data of trunk and affected hand will be recorded during subject imitations and will be analysed to assess any improvements.
Change in Oxford Cognitive Screen between two time points | Baseline and week 4
  is a stroke-specific cognitive screen

SECONDARY OUTCOMES:
Applicability perception and satisfaction degree of the proposed treatment | At week 4
  self-report questionnaire using a 5 point Likert scale (1 - Strongly disagree; 5 - Strongly agree). Higher score indicates greater satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Fadiga, MD, PhD, Study Director — Section of Human Physiology, University of Ferrara (Ferrara, Italy); Sofia Straudi, MD, PhD, Principal Investigator — Department of Neuroscience and Rehabilitation, University Hospital of Ferrara (Ferrara, Italy); Thierry Pozzo, PhD, Principal Investigator — IIT; Istituto Italiano di Tecnologia
Locations (1):
- Sofia Straudi, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No